CLINICAL TRIAL: NCT00568477
Title: Prospective, Randomized, Open, 2-arm National Multi-center Study to Evaluate the Value of Rituximab in Humoral Chronic Rejection After Renal Transplantation.
Brief Title: Value of Rituximab in Humoral Chronic Rejection After Renal Transplantation
Acronym: Rituximab 2006
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lacking recruitment
Sponsor: Technical University of Munich (Other)
Collaborators: Humboldt-Universität zu Berlin (Other); University of Erlangen-Nürnberg (Other); University Hospital, Essen (Other); University Hospital Freiburg (Other); Heidelberg University (Other); University of Jena (Other); Transplantationszentrum Köln-Merheim (Other); University of Regensburg (Other); Heinrich-Heine University, Duesseldorf (Other); Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Univ.-Prof. Dr. med. Dr. h.c. Uwe Heemann, Technical University of Munich, Klinikum rechts der Isar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAL-518-HEE-0200-S; EudraCT-number: 2006-006137-41
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2008-01

CONDITIONS: Grafting; Renal Transplantation; Transplantation, Kidney; Chronic Allograft Nephropathy
Keywords: Rituximab, Heemannn
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Treatment with rituximab
  Interventions: Drug: MabThera
- Arm 2 (No Intervention): Treatment without rituximab

INTERVENTIONS:
Drug: MabThera — Rituximab (MabThera):
  375 mg/m² as IV infusions over >=6h each at time point 0 and 2 weeks. Initial infusion rate of 50 mg/h, stepwise rise is possible after 30 minutes
  Arms: Arm 1

SUMMARY:
To evaluate the benefit of rituximab in patients with CAN with histologically proven C4d deposits and/or plasma cell and/or B-Lymphocyte (CD20+ cells) infiltration of their grafts.

DETAILED DESCRIPTION:
This study is a prospective, randomized, open, 2-arm, national multi-center study to evaluate the value of rituximab in humoral chronic rejection after renal transplantation in approximately 150-200 patients (75-100 patients each group).

All biopsies will be analysed by Prof. Groene (Heidelberg) and the results immediately communicated to the central managing unit (Munich). Upon receipt, patients with biopsy proven CAN with C4d+ and/or plasma-cells and/or B-lymphocytes within the last 4 weeks before inclusion (centrally confirmed), fulfilling the inclusion/exclusion criteria, will be randomized 1:1 into one of the 2 groups:

Arm 1: Treatment with rituximab Arm 2: Treatment without rituximab Recruitment will last for approximately one year. All patients will be treated with baseline medication of Tacrolimus, MMF, steroids (optional, with same dose as given before study entry) and ACE-inhibitor or AT1-receptor-antagonist. A single dose of 100 mg Methylprednisolone i.v. will be given at baseline (day 0) in both groups (in the rituximab group 30 min before start of the rituximab infusion).

Each patient will be followed for 1 year within protocol, with study visits at 1,3,7 and 14 days (rituximab group), 3, 6 and 12 months followed by a follow-up period of 1 year with a study visit at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Renal allograft recipients at least 1 year after transplantation with GFR > 25 ml/min x 1,73m2 (MDRD)
* Single organ recipients of renal allograft
* Patients who have provided informed consent
* Patients who are >= 18 years of age
* Patients who have biopsy proven CAN with C4d+ deposits and/or plasma-cells and/or B-lymphocytes within the last 4 weeks before inclusion
* Patients who are treated with ACE/AT1 Blocker more than 1 week before inclusion

Exclusion Criteria:

* Patients who suffer from HIV infection
* Patients with a history of Hepatitis B
* Patients with Hepatitis C (active/chronic)
* Patients who have a contraindication for the use of rituximab, such as leukopenia or experienced infusion-related adverse events to former antibody treatment
* Patients who showed signs of acute cellular rejection in the biopsy
* Patient has a malignancy or history of malignancy within the last 5 years, except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully.
* Patient has a systemic infection requiring treatment.
* Female patients who are pregnant or lactating
* Patients who have any form of substance abuse, psychological illness or any other condition, which, in the opinion of the investigator, may interfere with the patient's ability to understand the requirements of the study.
* Patients who have a proteinuria >4g/24h
* Patient is unlikely to comply with the visits scheduled in the protocol.
* Patient is simultaneously participating in another investigational drug study or has participated in such study within 28 days before entry in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-12; Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Primary objective: To evaluate the benefit of Rituximab in patients with CAN with histologically proven C4d deposits and/or B-Lymphocyte (CD20+ cells) infiltration of their grafts. Secondary objectives: Renal function at 1 year | Graft survival at 1 and 2 years

SECONDARY OUTCOMES:
Renal function at 1 year | Graft survival at 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Heemann, Prof. MD, Principal Investigator — Technical University of Munich, Klinikum rechts der Isar; Münchner Studienzentrum
Locations (1):
- Technical University of Munich, Munich, Bavaria, Germany